CLINICAL TRIAL: NCT07055802
Title: Effects Of Inversion Table Therapy Versus Mulligan Techniques On Pain And Lumbar Flexibility In Patients With Chronic Low Back Pain
Brief Title: Effects Of Inversion Table Therapy Vs MT On Pain And Lumbar Flexibility In Patients With Chronic Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/830
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inversion Table group (Experimental)
  Interventions: Combination Product: Inversion Table
- Mulligan group (Experimental)
  Interventions: Combination Product: Mulligan flexion biased exercises

INTERVENTIONS:
Combination Product: Inversion Table — Inversion Table group will receive flexion biased exercises in supine position with 05 repetitions every session and in addition will be given an inversion table therapy as a treatment at the angle of 60' for 5 minutes in every session. Two follow ups in a week were taken for total of 04 weeks. Measurements were taken for NPRS, Oswestry low back disability questionnaire and sit and reach test respectively
  Arms: Inversion Table group
Combination Product: Mulligan flexion biased exercises — experimental group named as Mulligan group will receive flexion biased exercises in supine position with 05 repetitions every session and in addition will be given mulligan technique. It was done at level just below ASIS (at level of L4-L5 spinous process), ten times/session, for 12 sessions three/week every other day for 4 weeks. . Measurements were taken for NPRS, Oswestry low back disability questionnaire and sit and reach test respectively
  Arms: Mulligan group

SUMMARY:
Chronic low back pain (CLBP) is a widespread yet difficult-to-manage and treat public health condition with a significant treatment failure rate. Both inversion table therapy and mulligan techniques are very effective in reducing low back pain. A number of literature supports the effectiveness of both techniques individually but there is no literature available that provide comparison between these two techniques.

DETAILED DESCRIPTION:
Study objective will be to compare the effect of inversion table therapy versus mulligan techniques on pain and lumber flexibility in patients with chronic low back pain

ELIGIBILITY:
Inclusion Criteria:

* Both Genders.
* Adults aged between 30-50.
* Low Back pain should be Persistent for more than 3 months
* Idiopathic pain

Exclusion Criteria:

* Pregnant females
* Patients with cauda equina syndrome (symptoms of bladder impairments)
* Cardiovascular disease in last 6 months
* Any progressive neurological deficit (like stroke and epilepsy)
* Patients history of vertigo and glaucoma
* Patient with flexion biased pain Persistent use of pain medication
* Patients who had undergone any other treatments, such as acupuncture or physical therapy, in last 3 months.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | 12 Months
  Oswestry disability index is used to identify level of disability or severity of lower back pain(20). For those suffering from low back pain (LBP), the Oswestry Disability Index is a commonly used outcome measure. It takes five minutes to complete and one minute to rate the self-administered ODI questionnaire. Scores correspond to a range of disabilities, from mild to bedridden. Time period for again filling of Oswestry questionnaire is 4 weeks. It is important to measure disability level in lower back pain and ODI is an important reliable tool to measure lower back disability. There are different scoring levels in percentage which indicates level of disability in ODI. From 0 to 4, there is no disability; from 5 to 14, a mild disability; from 15 to 24, a moderate disability; from 25 to 34, a severe disability; and from 35 to 50, a totally crippled person.
RAND SF-36 | 12 Months
  Rand SF-36 is a questionnaire used to assess quality of life. This tool consists of eight areas: physical function, vitality, emotional role function, general health awareness, physical aches, physical function, social function, and mental health. The higher the score, the better the quality of life. A score of 0 is equal to the maximum dysfunction, and a score of 100 means no dysfunction.
Sit and Reach Test | 12 Months
  Sit and Reach test is used to measure lumber flexibility through flexing lumber spine. In this test subject is in sitting position with legs fully extended and relaxed knee. Subject is asked to reach his arms as far as possible at flexibility meter and hold for 2 seconds. It comprises of different scores in cm categorised as 9 (very poor), 13 (poor), 14 (average), 15 (good), 17 (very good) and 25+ (excellent) Sit and reach test is found to be more reliable tool for measuring flexibility

CONTACTS AND LOCATIONS:
Locations (1):
- Omer Hospital & Cardiac Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No